CLINICAL TRIAL: NCT01394159
Title: Randomized Trial Comparing the 22-gauge Aspiration and 22-gauge Biopsy Needles for EUS-guided Sampling of Solid Pancreatic Mass Lesions
Brief Title: 22G FNA Needle vs. 22G ProCore Needle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: F110506010
Record Dates: First submitted 2011-07-12; First posted 2011-07-14 (Estimated); Results first posted 2015-04-01 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-02

CONDITIONS: Pancreatic Neoplasm
Keywords: passes required to establish diagnosis
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 22G ProCore biopsy needle (Active Comparator): Using the 22G ProCore needle for sampling pancreatic mass lesions, the tissue obtained will be compared to the standard FNA needle.
  Interventions: Procedure: 22G ProCore biopsy needle
- 22G standard FNA needle (Active Comparator): Using the 22G standard fine needle aspiration needle (FNA) for sampling pancreatic mass lesions, the tissue obtained will be compared to the 22 G ProCore needle.
  Interventions: Procedure: 22G standard FNA needle

INTERVENTIONS:
Procedure: 22G ProCore biopsy needle — Tissue will be acquired with the 22G Procore biopsy needle and the sample will be compared to the sample obtained with the 22G standard FNA needle.
  Other Names: Biopsy
  Arms: 22G ProCore biopsy needle
Procedure: 22G standard FNA needle — Tissue will be acquired with the 22G standard FNA biopsy needle and the sample will be compared to the sample obtained with the 22G ProCore biopsy needle.
  Other Names: biopsy
  Arms: 22G standard FNA needle

SUMMARY:
The aim of this research study is to identify the best needle for performing biopsy during EUS procedures. There are two types of needles for performing biopsy: A FNA needle that provides a small sample of tissue for analysis and a 22G ProCore needle that provides larger amount of tissue. It is not clear at this point which of the two needles is superior for performing biopsy. This study will attempt to identify the better needle by assessing the performance of both needles in a randomized fashion.

DETAILED DESCRIPTION:
In this randomized trial, the 22G standard fine needle aspiration needle was compared with the newly developed 22G ProCore needle for sampling pancreatic mass lesions during endoscopic ultrasound. Patients were randomized into the two needle groups and then various outcomes were compared between the two needle types, including the number of passes needed to establish a diagnosis, the ability to procure enough tissue sample to be able to make a diagnosis, the rates of needle failure and complication rates.

ELIGIBILITY:
Inclusion Criteria:

-All patients with solid pancreatic mass lesions

Exclusion Criteria:

* Coaguloapthy,
* minors,
* prgenant patients

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-07; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shyam Varadarajulu, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bang JY, Hebert-Magee S, Trevino J, Ramesh J, Varadarajulu S. Randomized trial comparing the 22-gauge aspiration and 22-gauge biopsy needles for EUS-guided sampling of solid pancreatic mass lesions. Gastrointest Endosc. 2012 Aug;76(2):321-7. doi: 10.1016/j.gie.2012.03.1392. Epub 2012 May 31. PMID 22658389

RESULTS

PARTICIPANT FLOW:
Groups:
- 22G ProCore Biopsy: Acquire biopsy with procore needle
  Procore Biopsy: Acquire tissue with procore biopsy needle
- 22G FNA Needle: Acquire tissue with 22 gauge fine needle aspiration needle
Period: Overall Study
Arm/Group | 22G ProCore Biopsy | 22G FNA Needle
Started | 28 | 28
Completed | 28 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ProCore Biopsy: Acquire biopsy with procore needle
  Procore Biopsy: Acquire tissue with procore biopsy needle
- FNA Needle: FNA: Acquire tissue with FNA needle
- Total: Total of all reporting groups
Arm/Group | ProCore Biopsy | FNA Needle | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (15.4) | 65.4 (11.1) | 65.2 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 15 | 16 | 31
Race/Ethnicity, Customized [Number; unit: participants]
  White | 22 | 21 | 43
  Black | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  United States | 28 | 28 | 56

OUTCOME MEASURES:

1. Primary Outcome: Compare the Median Number of Passes Required to Establish a Diagnosis
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: No. of passes for diagnosis
Arm/Group | 22G ProCore Biopsy | 22G FNA Needle
Number analyzed (Participants) | 28 | 28
No. of passes for diagnosis | 1 [1 to 1] | 1 [1 to 2.5]

2. Secondary Outcome: Diagnosis Achieved With the Needle
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | 22G ProCore Biopsy | 22G FNA Needle
Number analyzed (Participants) | 28 | 28
participants | 25 | 28

3. Secondary Outcome: Technical Failure
Description: Malfunction of the needle during endoscopic ultrasound-guided sampling of the pancreatic mass lesion before a diagnosis is achieved
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | 22G ProCore Biopsy | 22G FNA Needle
Number analyzed (Participants) | 28 | 28
participants | 1 | 0

ADVERSE EVENTS:
Arm/Group | 22G ProCore Biopsy | 22G FNA Needle
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 1/28 | 1/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 22G ProCore Biopsy (N=28) | 22G FNA Needle (N=28)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — This patient was in the FNA group and was managed conservatively
Mild acute pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — This patient was managed conservatively

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No